CLINICAL TRIAL: NCT05226026
Title: Impact of Improving Sleep and Reducing Opioid Use in Individuals With Chronic Pain on Central Pain Processing
Brief Title: NiteCAPP_HELPS_WD: Improving Sleep and Reducing Opioid Use in Chronic Pain Patients
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: NIDA R01 Awarded
Sponsor: University of Missouri-Columbia (Other)
Responsible Party: Principal Investigator, Christina McCrae, Professor, Director MizZzou Sleep Research Lab, University of Missouri-Columbia
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 2053802
Record Dates: First submitted 2021-11-08; First posted 2022-02-07 (Actual); Last update posted 2024-08-05 (Actual); Status verified 2024-08

CONDITIONS: Chronic Pain; Chronic Insomnia; Opioid Use
Keywords: Tapered withdrawal; NiteCAPP
MeSH Terms: conditions — Chronic Pain; Sleep Initiation and Maintenance Disorders

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- NiteCAPP HELPS (Experimental): 4 weeks of online CBT-I (1 session/week for 1 hour), followed by tapered withdrawal and motivational interviewing and check-ins.
  Interventions: Behavioral: NiteCAPP HELPS; Other: Tapered Withdrawal
- Treatment as Usual (Other): Continuation of standard treatment for sleep and pain for 4 weeks, followed by tapered withdrawal and motivational interviewing and check-ins.
  Interventions: Other: Tapered Withdrawal

INTERVENTIONS:
Behavioral: NiteCAPP HELPS — 4 weeks of NiteCAPP (a digital version of CBT-I recently developed at Mizzou)
  Arms: NiteCAPP HELPS
Other: Tapered Withdrawal — Gradual tapered withdrawal following CDC guidelines, with additional check-ins and motivational interviewing with a therapist.

SUMMARY:
This project addresses the highly significant problem of developing effective strategies for facilitating withdrawal from opioid medications. The proposed work is conceptualized within the context of a well-known theoretical framework (Cognitive Activation Theory of Stress), and the research questions are theory-driven. The team proposes to evaluate an innovative web-based version of CBT-I followed by tapered withdrawal in a randomized trial in comparison to a Treatment As Usual control followed by tapered withdrawal. The dependent measures have been well-selected to effectively evaluate the outcomes. The methodological details are rigorous.

DETAILED DESCRIPTION:
Individuals with chronic widespread pain are often prescribed opioid therapy. Unfortunately, opioid therapy offers questionable benefit for long-term pain management and is associated with other negative outcomes (arrhythmias, overdose, death). Individuals with chronic pain experience high rates of comorbid chronic insomnia, increased cognitive and physiological arousal, and disrupted executive function. They also often develop abnormal brain activation at rest and in response to painful stimuli (aka central sensitization). The investigator's research and other research shows individuals with chronic pain exhibit increased brain activation in the default mode network at rest and in regions associated with pain modulation in response to painful stimuli compared to healthy controls. Withdrawal from opioids can be difficult; and inadequately managed pain, abnormal brain activation, disrupted executive function, increased arousal, and poor sleep contribute to that difficulty. Consistent with the Cognitive Activation Theory of Stress (CATS), The investigators hypothesize that poor sleep and sustained arousal lead to critical changes in brain activation and disrupted executive function that increase pain and lead to opioid use. The proposed pilot will randomize 26 prescription opioid users who have chronic widespread pain and insomnia to 4 weeks of NiteCAPP (a digital version of CBT-I recently developed at Mizzou) or treatment as usual. They will then complete a gradual tapered withdrawal protocol for opioids.

ELIGIBILITY:
Inclusion Criteria:

* 18+ yrs old
* willing to be randomized
* can read/understand English
* diagnosed with chronic widespread pain and insomnia
* prescribed opioid medication for 1+ mo, 3+ times per week
* desire to reduce or eliminate opioid use
* written agreement from physician prescribing opioid medication
* no prescribed or OTC sleep meds for 1+ mo, or stabilized for 6+ wks.

Exclusion Criteria:

* unable to provide informed consent
* cognitive impairment (MMSE <26)
* sleep disorder other than insomnia [i.e., sleep apnea (apnea/hypopnea index, AHI >15), Periodic Limb Movement Disorder (myoclonus arousals per hour >15)]
* bipolar or seizure disorder (due to risk of sleep restriction treatment)
* other severe, untreated major psychopathology except depression or anxiety (e.g., suicidal ideation/intent, psychotic disorders)
* psychotropic or other medications (e.g., beta-blockers) that alter pain or sleep (medications prescribed for pain or sleep are allowed)
* participation in other non-pharmacological treatment for pain, sleep, or mood outside current Internal metal objects or electrical devices
* pregnancy
* presumptive/confirmed lumbar nerve root compression
* confirmed lumbar spinal stenosis
* <6 mos post back surgery
* other spinal disorders

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2022-03-31 (Actual); Primary Completion 2024-06-01 (Actual); Study Completion 2024-06-01 (Actual)

PRIMARY OUTCOMES:
Change in Insomnia Severity Index | Single administration at baseline, 8 weeks, following completion of gradual tapered withdrawal
  Insomnia severity; score range 0-28 (low severity - high severity)
Change in Pain Intensity - Daily Electronic Sleep Diaries | Single administration at baseline, 8 weeks, following completion of gradual tapered withdrawal
  Daily electronic dairies will record pain unpleasantness; range: 0-100 (none- most unpleasantness)
Change in Wake After Sleep Onset - Daily Electronic Sleep Diaries | Single administration at baseline, 8 weeks, following completion of gradual tapered withdrawal
  Daily electronic dairies will record wake after sleep onset (number of minutes)
Change in Sleep Onset Latency- Daily Electronic Sleep Diaries | Single administration at baseline, 8 weeks, following completion of gradual tapered withdrawal
  Daily electronic dairies will record sleep onset latency (number of minutes)
Change in Sleep Efficiency- Daily Electronic Sleep Diaries | Single administration at baseline, 8 weeks, following completion of gradual tapered withdrawal
  Daily electronic dairies will record sleep efficiency
Change in Fatigue - Daily Electronic Sleep Diaries | Single administration at baseline, 8 weeks, following completion of gradual tapered withdrawal
  Daily electronic dairies will record insomnia severity; range: 0-100 (no insomnia - most severe)
Change in Sleep and Pain Medication - Daily Electronic Sleep Diaries | Single administration at baseline, 8 weeks, following completion of gradual tapered withdrawal
  Daily electronic dairies will record daily medication consumption
Change in Perceived Stress Scale | Single administration at baseline, 8 weeks, following completion of gradual tapered withdrawal
  Perception of stress; score range: 0-40 (low stress - high stress)
Change in Peripheral Arousal | 5 mins at rest at baseline, 8 weeks, following completion of gradual tapered withdrawal
  Heart Rate Variability (as measured by Holter-Monitoring)
Change in Pain Catastrophizing Scale | Single administration at baseline, 8 weeks, following completion of gradual tapered withdrawal
  The PCS yields a total score and three subscale scores assessing rumination, magnification and helplessness. Total score range from 0-52, with higher scores indicating greater pain catastrophizing.
Change in Neural Imaging: Structural/Functional MRI/Diffusion Weighted Imaging | Single administration at baseline, 8 weeks, following completion of gradual tapered withdrawal
  assessment of neural plasticity
Change in Thermal Pain Response | Single administration at baseline, 8 weeks, following completion of gradual tapered withdrawal
  Participants will undergo quantitative sensory testing using a contact thermode applied to the left plantar, VAS scale for pain ()-100)
Change in Opioid Use (Quantitative) | Single administration at baseline, 8 weeks, following completion of gradual tapered withdrawal
  Change in opioid use assessed with quantitative urine opioid panel
Change in Opioid Use (Self-Report) | Single administration at baseline, 8 weeks, following completion of gradual tapered withdrawal
  Change in opioid use assessed with daily electronic diaries

SECONDARY OUTCOMES:
Change in State-Trait Anxiety Inventory (STAI) | Single administration at baseline, 8 weeks, following completion of gradual tapered withdrawal
  Trait and state anxiety; score range: 20-80 (low anxiety - high anxiety)
Change in Depression (Beck Depression Inventory-II) | Single administration at baseline, 8 weeks, following completion of gradual tapered withdrawal
  Depression severity; score range: 0-63 (normal - extreme depression)
Change in 36-Item Short Form Survey (SF-36) | Single administration at baseline, 8 weeks, following completion of gradual tapered withdrawal
  Self-reported health; score range: low quality of life to high quality of life
Change in Objective Wake After Sleep Onset (Actigraph) | Single administration at baseline, 8 weeks, following completion of gradual tapered withdrawal
  Wake after sleep onset via Actiwatch-2
Change in Objective Sleep Onset Latency (Actigraph) | Single administration at baseline, 8 weeks, following completion of gradual tapered withdrawal
  Sleep Onset Latency via Actiwatch-2
Change in Objective Sleep Efficiently (Actigraph) | Single administration at baseline, 8 weeks, following completion of gradual tapered withdrawal
  Sleep Efficiency via Actiwatch-2
Change in NIH Toolbox | Single administration at baseline, 8 weeks, following completion of gradual tapered withdrawal
  20 minute computerized cognitive tasks
Change in non-opioid substance use | Single administration at baseline, 8 weeks, following completion of gradual tapered withdrawal
  self reported changes in non-opioid substances via electronic diaries

OTHER OUTCOMES:
Satisfaction Survey | Single administration at post-treatment - 8 weeks, following completion of gradual tapered withdrawal
  Experience with the assessments, procedures, and other features of the research study; score range: 9-90 (low satisfaction - high satisfaction)

CONTACTS AND LOCATIONS:
Locations (1):
- University of Missouri-Columbia, Columbia, Missouri, United States

IPD SHARING:
Plan to Share IPD: No